CLINICAL TRIAL: NCT01055548
Title: Parents Views on Diagnosis and Information-giving in Neonatal Care (Pilot Study)
Brief Title: PPrime: Parents Views on Diagnosis and Information-giving in Neonatal Care (Pilot Study)
Acronym: PPrime
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: EudraCT 2009-0138888-19
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2010-01

CONDITIONS: Parents of Preterm Infants Born Before 33 Weeks Gestation
Keywords: Preterm; Perinatal; Ultrasound; Cerebral palsy; Anxiety; Parents
MeSH Terms: conditions — Premature Birth; Cerebral Palsy; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Parents of babies born before 33 weeks gestation

SUMMARY:
The aim of the pilot study is to explore and identify the issues of concern to parents whose babies have been cared for in a neonatal unit and exposed to imaging, its influence on diagnosis and information-giving process

DETAILED DESCRIPTION:
The aim is to explore the recent experience and views of parents in a qualitative way to assist the development of a questionnaire which can be used with a much larger group of parents. The interview guide with the topics to be covered will include: expectations, concerns and issues relating to the equipment used with their baby, any investigations, including cranial ultrasound and MR imaging and the information provided.

The data collected will then inform the development of a standard instrument or questionnaire which will be used with parents participating in a trial using a randomised design to compare the influence of MR and ultrasound-based information on parental perceptions, stress and coping in association with healthcare usage and costs.

ELIGIBILITY:
Inclusion Criteria:

* Parents of babies born before 33 weeks gestation Parents who are 16 years of age or older Parents who are able to give informed consent Parents who are able to take part in interviews which are conducted in English

Exclusion Criteria:

* Parents who are under 16 years of age Parents who are unable to give informed consent Parents who are unable to take part in interviews which are conducted in English Parents where there are possible or know child protection issues

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents of babies born before 33 week's gestation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor D Edwards, Principal Investigator — Imperial College London; Dr D Azzopardi, Principal Investigator — Imperial College London; Dr M Redshaw, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, United Kingdom